CLINICAL TRIAL: NCT00392210
Title: Assessment of Two Postoperative Techniques Used to Predict Voiding Efficiency After Gynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 15107
Record Dates: First submitted 2006-10-23; First posted 2006-10-25 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spontaneous Fill (No Intervention)
- Retrograde Fill (Active Comparator)
  Interventions: Genetic: Voiding Trial

INTERVENTIONS:
Genetic: Voiding Trial — Post-void residual and uroflow study will be done twice
  Arms: Retrograde Fill

SUMMARY:
After gynecologic surgery, it may be difficult to void (urinate). This problem is usually short-term with normal function returning within a few days to a few weeks. For this reason, patients may require drainage of their bladder with a catheter immediately after surgery. Currently in our office, we use two different tests to see how well you are able to urinate and how quickly the catheter can be removed. The purpose of this study is to see which voiding test is better after gynecologic surgery.

DETAILED DESCRIPTION:
Postoperative voiding dysfunction is commonly encountered following gynecologic surgery. This dysfunction is usually short term, with normal function returning within a few days. Following uro/gynecologic surgery, most patients require drainage with either a transurethral or suprapubic catheter in the immediate postoperative period. Within our practice, we prefer drainage with a transurethral catheter.

At some point after surgery, the urethral catheter is removed and normal bladder function allowed to resume. At present, there is no generally accepted regimen to assess voiding efficiency. In our practice, we currently employ two regimens to both assess voiding efficiency and expedite catheter removal. In one technique, the catheter is removed and the patient's bladder is allowed to fill spontaneously. Patients are asked to void when they experience a strong urge. The voided volume is recorded and a post-void residual (PVR) is then measured by transurethral straight catheterization.

In the second technique, the patient's bladder is retrogradely filled with 300 cc of sterile fluid and the catheter removed. They are asked to void within 15 minutes of instillation and the voided volume is measured. The PVR is then obtained by transurethral straight catheterization.

In both cases, if the patient voids >2/3 the total volume (voided volume + residual) the trial is considered "passed" and the catheter is removed. If a patient voids < 2/3 of the total volume, the trial is considered "failed" and indicative of urinary retention. In this case the catheter replaced.

We aim to assess the ability of these techniques to accurately predict voiding efficiency and to determine if one technique is superior to the other.

ELIGIBILITY:
Inclusion Criteria:

* All women > 18 years of age presenting to the Division of Urogynecology at the University of Rochester Medical Center/Strong Memorial Hospital and undergoing gynecologic surgery which requires postoperative placement of a transurethral catheter.
* Subjects must be competent to give informed consent.

Exclusion Criteria:

* Any patient less than 18 years of age.
* Patients with suprapubic catheters postoperatively.
* Patients undergoing surgery that does not require transurethral catheterization postoperatively.
* Patients not competent to give informed consent.
* Patients who are pregnant.
* Patients undergoing procedures requiring prolonged bladder decompression (i.e. fistula repair).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael K. Flynn, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 271 potential subjects were identified. 192 declined participation so 79 were enrolled.
Pre-assignment Details: 10 subjects were withdrawn prior to randomization
Groups:
- Auto-fill Followed by Back Fill: The Auto fill-method was performed immediately followed by the back-fill method. Auto fill: The catheter was removed and the bladder was allowed to fill spontaneously until the patient experienced a strong urge to void. Back Fill: The bladder was filled retrograde through the indwelling Foley catheter with 300 cc sterile saline or until the patient reported a strong urge whichever occurred first.
- Back Fill Followed by Autofill: The back fill-method was performed immediately followed by the auto-fill method. Auto fill: The catheter was removed and the bladder was allowed to fill spontaneously until the patient experienced a strong urge to void. Back Fill: The bladder was filled retrograde through the indwelling Foley catheter with 300 cc sterile saline or until the patient reported a strong urge whichever occurred first.
Period: First Voiding Trial
Arm/Group | Auto-fill Followed by Back Fill | Back Fill Followed by Autofill
Started | 36 | 33
Completed | 34 | 31
Not Completed | 2 | 2
Not completed — Physician Decision | 2 | 2
Period: Second Voiding Trial
Arm/Group | Auto-fill Followed by Back Fill | Back Fill Followed by Autofill
Started | 34 | 31
Completed | 34 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Auto Fill Followed by Back Fill: The Auto fill-method was performed immediately followed by the back-fill method. Auto fill: The catheter was removed and the bladder was allowed to fill spontaneously until the patient experienced a strong urge to void. Back Fill: The bladder was filled retrograde through the indwelling Foley catheter with 300 cc sterile saline or until the patient reported a strong urge whichever occurred first.
- Back Fill Followed by Auto Fill: The back fill-method was performed immediately followed by the auto-fill method. Auto fill: The catheter was removed and the bladder was allowed to fill spontaneously until the patient experienced a strong urge to void. Back Fill: The bladder was filled retrograde through the indwelling Foley catheter with 300 cc sterile saline or until the patient reported a strong urge whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Auto Fill Followed by Back Fill | Back Fill Followed by Auto Fill | Total
Number analyzed (Participants) | 41 | 38 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 21 | 46
  >=65 years | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.73 (12.05) | 57.58 (10.04) | 59.02 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 38 | 79
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 38 | 79

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Passed Bladder Trial
Description: Voiding trial 1 was performed according to the patient assignment to group 1 or 2. Voiding trial 2 was done immediately after completion of trial 1. A successful trial was defined as a void of greater than two-thirds of total bladder volume (voided volume + post-void residual urine).
Time Frame: postoperatively after surgery on day1 or 2
Measure: Number; unit: participants
Groups:
- Auto Fill Intervention: Auto fill: The catheter was removed and the bladder was allowed to fill spontaneously until the patient experienced a strong urge to void.
- Back Fill Intervention: Back Fill: The bladder was filled retrograde through the indwelling Foley catheter with 300 cc sterile saline or until the patient reported a strong urge whichever occurred first.
Arm/Group | Auto Fill Intervention | Back Fill Intervention
Number analyzed (Participants) | 65 | 65
participants | 25 | 39

ADVERSE EVENTS:
Groups:
- Auto Fill: Auto fill: The catheter was removed and the bladder was allowed to fill spontaneously until the patient experienced a strong urge to void.
- Back Fill: Back Fill: The bladder was filled retrograde through the indwelling Foley catheter with 300 cc sterile saline or until the patient reported a strong urge whichever occurred first.
Arm/Group | Auto Fill | Back Fill
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/69
Other Adverse Events (participants affected / at risk) | 0/69 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No